CLINICAL TRIAL: NCT00889590
Title: Adjuvant Zoledronic Acid in 'High Risk' Giant Cell Tumour of Bone (GCT) - A Randomized Phase II Study
Brief Title: Adjuvant Zoledronic Acid in High Risk Giant Cell Tumour of Bone (GCT)
Acronym: HR-GCT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment with registration denosumab
Sponsor: Leiden University Medical Center (Other)
Responsible Party: Principal Investigator, J.R. Kroep, MD PhD, Leiden University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P08.185
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Giant Cell Tumor of Bone; Osteoclastoma
Keywords: GCT; Bisfosfonates
MeSH Terms: conditions — Giant Cell Tumor of Bone | interventions — Zoledronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Zoledronic acid (Experimental): Adjuvant zoledronic acid
  Interventions: Drug: Zoledronic acid
- Control (No Intervention): Standard care

INTERVENTIONS:
Drug: Zoledronic acid — 4 mg, monthly for 3 months followed by a 3-monthly schedule for up to one year after surgery
  Other Names: Zometa
  Arms: Zoledronic acid

SUMMARY:
This is a multicenter, randomised phase II trial in patients with high risk GCT.

Primary objective:

* Determine if adjuvant zoledronic acid improves the 2 years recurrence rate of 'high risk' GCT as compared to standard care

Secondary objectives:

* Determine the relapse free survival
* Evaluate the usefulness of bone remodelling markers in diagnosing and monitoring GCT

DETAILED DESCRIPTION:
GCT is a potentially malignant tumour that presents with a locally destructive osteolytic lesion. The high risk GCT are characterized by a high recurrence rate around the 40-45%. Zoledronic acid is a potent inhibitor of osteolysis and is capable of inducing osteoclast and stromal cell apoptosis, which makes it an attractive adjuvant treatment in 'high risk' GCT in order to improve clinical outcomes and reduce the recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male or female > 18 years of age
* Histologically proven GCT treated with surgery
* High risk GCT defined as minimal one or more of the following:

  * Recurrent GCT
  * GCT located in the pelvis, sacrum, spine, distal ulna or growth in soft tissue
  * GCT grade III
  * Pathological fracture in GCT
  * Absence of local adjuvant therapy (cryosurgery or phenol instillation)
* Neutrophils > 1.5x109/L, platelets > 100x109/L, and Hb > 6 mmol/l
* Bilirubin level < 1.5 x ULN
* ASAT and ALAT < 2.5 x ULN
* Adequate renal function as defined by: serum creatinine clearance > 60 cc/min
* Expected adequacy of follow-up

Exclusion Criteria:

* Unresectable or metastatic GCT and grade IV GCT
* Prior bisphosphonate usage, except preoperative treatment with zoledronic acid up to 3 months before surgery
* Other previous malignancy within 5 years, with exception of a history of a previous basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Known hypersensitivity reaction to any of the components of the treatment
* Pregnancy or lactating
* Medical or psychological condition which in the opinion of the investigator would not permit the patient to complete the study or sign meaningful informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-12; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Determine if adjuvant zoledronic acid improves the 2 year recurrence rate of 'high risk' GCT as compared to standard care | 4 years

SECONDARY OUTCOMES:
Evaluate the usefulness of bone remodelling markers in diagnosing and monitoring GCT | 4 years
Determine the relapse free survival | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: J R Kroep, MD PhD, Principal Investigator — Leiden University Medical Center (LUMC); P D Dijkstra, MD PhD, Study Director — LUMC; A H Taminiau, MD PhD, Study Director — LUMC; P C Hogendoorn, MD PhD, Study Director — LUMC; H Gelderblom, MD PhD, Study Director — LUMC; N A Hamdy, MD PhD, Study Director — LUMC; S E Papapoulos, MD PhD, Study Director — LUMC
Locations (4):
- University hospital Gent, Ghent, Belgium
- Netherlands (3):
  - Academic Medical Center, University of Amsterdam, Amsterdam
  - Groningen University Medical Center, Groningen
  - Leiden University Medical Center, Leiden

REFERENCES:
- [Derived] Lipplaa A, Kroep JR, van der Heijden L, Jutte PC, Hogendoorn PCW, Dijkstra S, Gelderblom H. Adjuvant Zoledronic Acid in High-Risk Giant Cell Tumor of Bone: A Multicenter Randomized Phase II Trial. Oncologist. 2019 Jul;24(7):889-e421. doi: 10.1634/theoncologist.2019-0280. Epub 2019 Apr 30. PMID 31040253